CLINICAL TRIAL: NCT01791829
Title: A Prospective Cohort Study Evaluating Risk of Local Recurrence Following Breast Conserving Surgery and Endocrine Therapy in Low Risk Luminal A Breast Cancer
Acronym: LUMINA
Status: Active, not recruiting | Type: Observational
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: OCOG-2012-LUMINA
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Luminal A; Ipsilateral Breast Tumour Recurrence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be used to determine Ki67 status by IHC and subsequent testing for DNA/RNA.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Luminal A with other Clinical Criteria: BCS postulated to be at low risk for IBTR following Endocrine Therapy

SUMMARY:
This is a multicentre, single-arm prospective cohort study evaluating risk of ipsilateral breast tumour recurrence(IBTR) following breast conserving surgery (BCS) in a group of women postulated to be at low risk for recurrence. Women with luminal A breast cancer determined by immunohistochemical(IHC) and other low risk clinical testing (see below) will be treated with endocrine therapy (tamoxifen or aromatase inhibitor) for five years and will not be treated with breast irradiation (BI). Subjects will be followed for 10 years and will be assessed for recurrent disease, new primary cancer and survival.

DETAILED DESCRIPTION:
The independent prognostic ability of the luminal A subtype has been demonstrated in two retrospective analyses of prospective trials and suggests that luminal A combined with other known clinical prognostic factors could be used to select patients treated with BCS at very low risk for IBTR who could avoid BI. Given that using intrinsic subtyping combined with other clinical factors to identify women who could avoid BI would be a major change in clinical practice, we propose that a prospective study is necessary to confirm that such an approach can accurately identify a group of women at very low risk for IBTR following BCS.

We anticipate that the risk of IBTR in the low risk group is likely to be lower than that observed in previous trials (predicted to be < 5% at 5 years and < 10% at 10 years) for several reasons: first, our selection criteria (node negative, luminal A, > or = 55 years, tumours < or = 2cm, excision margin > or = 1mm post-BCS, absence of lobular cancers, extensive intraductal component and lymphovascular invasion) are more restrictive than in previous trials and second, the risks of IBTR are steadily decreasing over time due to improvements in mammographic screening, pre-op staging, tumour localization, and surgical practice. The expected low failure rates are unlikely to warrant the use of radiation.

A prospective cohort study was identified as the most appropriate and efficient design as our primary hypothesis is that a group of patients at very low risk of IBTR can be identified. A randomized trial could address the effectiveness of radiation in such a cohort of patients, but would require a much larger sample size to detect very small differences, which would not be clinically meaningful. During the conduct of this trial it is anticipated that patients who do not meet study criteria or who decline study enrollment, will continue to receive BI after BCS.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient > or = 55 years of age with a new diagnosis of invasive carcinoma of the breast (ductal, tubular or mucinous only) with primary tumour < or =2cm on microscopic exam, with no evidence of metastatic disease;
2. ER positive (> or =1%) and PR positive (>20%) and HER2 negative (Immunohistochemical (IHC) or In Situ Hybridization (ISH) approach);
3. Treated by BCS with microscopically clear resection margins > or = 1mm for invasive and non-invasive disease or no residual disease on re-excision;
4. Negative axillary node involvement determined by sentinel node biopsy or axillary node dissection.

Exclusion Criteria:

1. Clinical or pathological evidence of T4 disease (i.e. extension to chest wall, skin involvement, peau d'orange, or inflammatory breast cancer).
2. Multifocal or multicentric disease.
3. Evidence of an extensive intraductal component (defined as a tumour that is composed of 25% or more of DCIS and the DCIS extends beyond the gross dimensions of the tumour), or disease limited to micro invasion only.
4. Grade 3 histology for invasive disease
5. Evidence of lymphovascular invasion.
6. Evidence of disease on pre-operative mammogram, aside from primary cancer treated by breast conserving surgery.
7. Bilateral malignancy of the breast (synchronous or metachronous).
8. Known BRCA 1 or 2 mutations.
9. History of non-breast cancer malignancies if not disease free for > 5 years and considered low risk of recurrence with the exception of treated carcinoma in-situ of the cervix, endometrium or colon, melanoma in-situ and basal or squamous cell carcinoma of the skin.
10. Serious non-malignant disease associated with a life expectancy < 10 years.
11. Inability to be treated with or to tolerate endocrine therapy.
12. Psychiatric or addictive disorder, which would preclude obtaining informed consent or adherence to protocol.
13. Geographic inaccessibility for follow-up.
14. Inability to understand or unable to provide written informed consent.
15. Inability to be registered on study within 12 weeks of the last surgical procedure on the breast.
16. Central testing for Ki67 > 13.25% consistent with the luminal B subtype

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicentre, single-arm prospective cohort study evaluating risk of IBTR following BCS in a group of women postulated to be at low risk for recurrence. Subjects will be followed for 10 years and will be assessed for recurrent disease, new primary cancer and survival. The primary outcome is IBTR
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral Breast Tumour Recurrence (IBTR) | 5 years
  The primary outcome is IBTR defined as recurrent invasive or in-situ cancer in the ipsilateral breast during follow-up. Histological evidence of recurrence will be required. All recurrences will be reviewed by a central adjudication committee.

SECONDARY OUTCOMES:
Recurrence Free interval (RFI) | 5 years
  Recurrence free interval (RFI) defined as time from registration to time of documented recurrent disease (ipsilateral breast, regional or distant)
Event-free survival (EFS) | 5 years
  Event-free survival (EFS) defined as the time from registration to the time of documented IBTR, regional (ipsilateral axilla, supraclavicular or internal mammary nodes), distant recurrence (bone, liver, lung, brain, etc.), contralateral breast cancer, new primary cancer or death
Overall survival (OS) | 5 years
  Overall survival (OS) defined as time from registration to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Tim Whelan, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG); Sally Smith, MD, Principal Investigator — British Columbia Cancer Agency (BCCA)
Locations (27):
- Canada (27):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Abbotsford Centre, Abbotsford, British Columbia
  - BC Cancer Agency, Centre for the North, Prince George, British Columbia
  - BCCA - Vancouver Centre, Vancouver, British Columbia
  - BC Cancer Agency, Victoria, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Centre, London, Ontario
  - R.S. McLaughlin Durham Regional Cancer Centre, Oshawa, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre integre de sante et de services sociaux de laval (CISSS de Laval), Laval, Quebec
  - CHUM - Hopital Notre Dame, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - CHUQ - Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - CHUS - Hopital Fleurimont, Sherbrooke, Quebec
  - The Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen TO, Leung SCY, Riaz N, Mulligan AM, Kos Z, Bane A, Whelan TJ. Ki67 assessment protocol as an integral biomarker for avoiding radiotherapy in the LUMINA breast cancer trial. Histopathology. 2023 Dec;83(6):903-911. doi: 10.1111/his.15032. Epub 2023 Aug 23. PMID 37609778
- [Derived] Whelan TJ, Smith S, Parpia S, Fyles AW, Bane A, Liu FF, Rakovitch E, Chang L, Stevens C, Bowen J, Provencher S, Theberge V, Mulligan AM, Kos Z, Akra MA, Voduc KD, Hijal T, Dayes IS, Pond G, Wright JR, Nielsen TO, Levine MN; LUMINA Study Investigators. Omitting Radiotherapy after Breast-Conserving Surgery in Luminal A Breast Cancer. N Engl J Med. 2023 Aug 17;389(7):612-619. doi: 10.1056/NEJMoa2302344. PMID 37585627
- See also: Related Info — http://www.ocog.ca